CLINICAL TRIAL: NCT04859764
Title: Effects of Corticosteroid Injection Plus Reparel™ Knee Sleeve on Knee Osteoarthritis: A Randomized Clinical Trial
Brief Title: Effect of Reparel Knee Sleeve With Knee Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Amit Momaya, Assistant Professor, Section Chief, Sports Medicine, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-300006118
Record Dates: First submitted 2021-03-02; First posted 2021-04-26 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Adrenal Cortex Hormones; Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unmarked sleeves will be used. Half will be Reparel sleeves, and half will be placebo. Participants and sleeve numbers will be randomized via REDCap.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Reparel Sleeve Group (Experimental): Reparel sleeve and corticosteroid injection
  Interventions: Device: Reparel knee sleeve; Drug: Corticosteroid injection
- Placebo Sleeve Group (Placebo Comparator): Placebo sleeve and corticosteroid injection
  Interventions: Drug: Corticosteroid injection; Device: Placebo knee sleeve

INTERVENTIONS:
Device: Reparel knee sleeve — Unlabelled thermo-active knee sleeve that improves bloodflow to knee and decreased pain
  Arms: Reparel Sleeve Group
Drug: Corticosteroid injection — intraarticular knee injection of betamethasone and bupivacaine 0.5% (dose is determined by joint size)
  Other Names: betamethasone and bupivacaine 0.5%
Device: Placebo knee sleeve — unlabeled compression knee sleeve
  Arms: Placebo Sleeve Group

SUMMARY:
The goals of treating knee osteoarthritis (OA) is to improve or maintain quality of life, mobility and function, pain relief, and improve inflammation. The different treatment options for knee OA have been extensively studied and implemented, but the optimum treatment is still undecided. There is a belief that anti-inflammatory sleeve technology may be beneficial in treating knee OA. The purpose of this study is to determine if the Reparel™ knee sleeve results in superior mobility, functionality, and pain outcomes as compared to a placebo knee sleeve in managing knee OA.

DETAILED DESCRIPTION:
Patients who are recommended non-operative management of their knee osteoarthritis and have consented to participate in the study will be randomized into two groups to receive either of the following

1. Reparel knee sleeve
2. Placebo knee sleeve

Participants assigned to both groups will be given instructions on how to use/wear the sleeve while performing activities of daily living or sports that had previously resulted in knee pain and also be asked to do the follows:

* Wear the sleeve as much as they possibly can
* Not change their usual activities and diet during the time they are on this study.
* Record in a diary the number of hours sleeve was worn per day
* Record any adverse effects or discomfort due to sleeve use.
* Not to receive any injections in the subsequent 6 months following baseline randomization visit.

Participant background information that is relevant to this study will also be collected from their medical record including age, sex, and race and stored in a hospital secure computer database (REDCap).

Participants will also be asked to complete the Knee Injury and Osteoarthritis Outcome Score (KOOS), Single Assessment Numeric Evaluation (SANE), Oxford Knee Score (OKS), Lysholm Score, UCLA Activity Score and Visual Analog Scale (VAS) survey questionnaires at baseline randomization visit (T0), at 4 weeks (T1), at 3 months (T2), and at 6 months (T3) to assess the mobility, functionality, and pain associated with the affected leg.

The responses to the surveys will be recorded on a password-protected laptop and all patient identifiers will be replaced with unique identifier numbers. Only the study team will have access to the responses from the forms. The analysis of de-identified data will be done through SPSS 27, and scores for the questionnaires will be averaged and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* osteoarthritis visible on knee radiograph
* patient opting for non-surgical treatment

Exclusion Criteria:

* bilateral symptomatic knee osteoarthritis
* prior surgery on the knee of interest
* hardware present on the knee of interest
* gross instability detected on physical exam
* malignancy in the knee of question

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Change in University of California, Los Angeles (UCLA) Activity Score at 4 weeks | 4 weeks (T1)
  activity score, 1-10, 10 is best outcome
Change in University of California, Los Angeles (UCLA) Activity Score at 3 months | 3 months (T2)
  activity score, 1-10, 10 is best outcome
Change in University of California, Los Angeles (UCLA) Activity Score at 6 months | 6 months (T3)
  activity score, 1-10, 10 is best outcome
Change in Lysholm Score at 4 weeks | 4 weeks (T1)
  ability to manage activities of daily living, 0-100, 100 is best outcome
Change in Lysholm Score at 3 months | 3 months (T2)
  ability to manage activities of daily living, 0-100, 100 is best outcome
Change in Lysholm Score at 6 months | 6 months (T3)
  ability to manage activities of daily living, 0-100, 100 is best outcome
Change in Oxford Knee Score (OKS) at 4 weeks | 4 weeks (T1)
  knee pain and function score, 0-48, 48 is best outcome
Change in Oxford Knee Score (OKS) at 3 months | 3 months (T2)
  knee pain and function score, 0-48, 48 is best outcome
Change in Oxford Knee Score (OKS) at 6 months | 6 months (T3)
  knee pain and function score, 0-48, 48 is best outcome
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 4 weeks | 4 weeks (T1)
  knee pain and function score, 0-100, 100 is best outcome
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 3 months | 3 months (T2)
  knee pain and function score, 0-100, 100 is best outcome
Change in Knee Injury and Osteoarthritis Outcome Score (KOOS) at 6 months | 6 months (T3)
  knee pain and function score, 0-100, 100 is best outcome
Change in Single Assessment Numeric Evaluation (SANE) at 4 weeks | 4 weeks (T1)
  function score, 0-100%, 100% is best outcome
Change in Single Assessment Numeric Evaluation (SANE) at 3 months | 3 months (T2)
  function score, 0-100%, 100% is best outcome
Change in Single Assessment Numeric Evaluation (SANE) at 6 months | 6 months (T3)
  function score, 0-100%, 100% is best outcome
Need for Additional CSI | 6 months
  need for additional CSI after baseline injection
Change in Visual Analog Scale (VAS) at 4 weeks | 4 weeks (T1)
  pain score, 0-10, 10 is best outcome
Change in Visual Analog Scale (VAS) at 3 months | 3 months (T2)
  pain score, 0-10, 10 is best outcome
Change in Visual Analog Scale (VAS) at 6 months | 6 months (T3)
  pain score, 0-10, 10 is best outcome

SECONDARY OUTCOMES:
Satisfaction with knee sleeve at 4 weeks | 4 weeks (T1)
  0-10, 10 is best
Satisfaction with knee sleeve at 3 months | 3 months (T2)
  0-10, 10 is best
Satisfaction with knee sleeve at 6 months | 6 months (T3)
  0-10, 10 is best
Average wear time of sleeve over past week at 4 weeks | 4 weeks (T1)
  0-24 hours, 24 hours is best
Average wear time of sleeve over past week at 3 months | 3 months (T2)
  0-24 hours, 24 hours is best
Average wear time of sleeve over past week at 6 months | 6 months (T3)
  0-24 hours, 24 hours is best

CONTACTS AND LOCATIONS:
Overall Officials: Amit Momaya, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Hospital Highlands, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No